CLINICAL TRIAL: NCT00971256
Title: Urine Cytology and Utility in Bladder Recurrence
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-144
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Bladder Cancer
Keywords: Bladder; Cancer; Cytology
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bladder cancer patients: Bladder cancer patients from one Beaumont Urologist.

SUMMARY:
Review bladder cancer patients and form a database in regards to urine cytology.

DETAILED DESCRIPTION:
In 2008 there was an estimated 68,810 new cases of bladder cancer, and 14,100 deaths. On the list of morbidity due to cancer, bladder cancer ranks number nine, yet is number one in dollars spent per cancer diagnosis and treatment.

Guidelines include cystoscopy and cytology/urine study every three months for the first 2 years and then every 6 months for the next 2 years, with the cycle being reset with every recurrence.

Urine cytology currently considered the gold standard for urine tests has many pros and cons. The points that keep it in use include: its high specificity, the ability to detect upper tract occurrence, and the ability to monitor the small population of those with bladder cancer whose disease becomes more aggressive. Opponents to cytology refer to the fact that is has low sensitivity that it is fairly subjective and that newer markers in comparison are improved.

There are multiple journal article which document the performance of cytology and the newer markers, the new markers versus cytology and then the performance of cytology in tandem with these new markers. The bottom line that is often overlooked is that cytology is expensive and each of the newer markers are at least as expensive as cytology. With the fact that a person who is diagnosed with non invasive bladder cancer can have up to 13 urine cytology's in 5 years without any recurrence we believe newer rational recommendations need to be made in regards to urine studies and bladder cancer follow up.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer patients from Dr. Jay Hollander's private practice.

Exclusion Criteria:

* Patients with diagnosis of bladder cancer without initial cytology available.
* Patients who received outside nephrectomy or cystectomy without pathology available.
* Those who had recurrence without cytology results available.
* Those who were followed by Dr Hollander and another urologist in which records are missing for a significant number of follow ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Review bladder cancer patients and form a database in regards to urine cytology. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mashni, MD, Principal Investigator — Beaumont Hospitals